CLINICAL TRIAL: NCT06032611
Title: Interest of Two Digital Devices for the Diagnosis of Neurocognitive Disorders in Elderly People With Cognitive Symptoms.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RIVAGES (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Université d'Évry (Other); Hôpital Charles Foix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: COGNUM; IDRCB2022-A00609-34 (Other: ANSM)
Record Dates: First submitted 2023-09-01; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Age-related Cognitive Decline; Computers, Handheld; Neurocognitive Disorders
Keywords: tablet; smartwatch; diagnosis
MeSH Terms: conditions — Neurocognitive Disorders; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will complete a number of cognitive and fine motor tests on a touch-sensitive tablet. They will also be asked to complete a questionnaire on their habits and medical history. They will also be asked to wear a smartwatch for 7 days.
  Interventions: Diagnostic Test: COGNUM_ALZVR

INTERVENTIONS:
Diagnostic Test: COGNUM_ALZVR — Participants will complete a battery of tests/quizzes:
  * cognitive tests
  * medical questionnaire
  * lifestyle/fragility questionnaire
  * digital clock test
  * fine motor skills tests They will also wear a connected watch for 7 days.

SUMMARY:
The goal of this clinical trial is to compare conventional clinical data collected as part of usual practice with data collected by the two digital tools to help diagnose major and minor neurocognitive disorders in elderly people consulting a memory center for cognitive complaints. The main question[s] it aims to answer are:

* Is it possible to create a classification between the different intensities of cognitive impairment?
* Is it possible to create a diagnostic tool consistent with the reference diagnosis? Participants will be asked to complete a series of cognitive and fine motor tasks, and will be given questionnaires on their lifestyle and medical history. They will be asked to wear a connected watch for 1 week.

There is no comparison group.

DETAILED DESCRIPTION:
Alzheimer's disease, which leads to dementia, has an insidious onset and a slow, gradual progression. After a completely asymptomatic phase that can last several years (prodromal stage of the disease), the first signs consist of a moderate deterioration in performance in one or more cognitive domains, such as memory, attention, planning or other cognitive faculties. Clinically, this is referred to as mild neurocognitive impairment (MCI) due to Alzheimer's disease. The progression is towards a major neurocognitive disorder, in which cognitive dysfunction progressively increases, and the patient becomes dependent for activities of daily living. Early detection of the disease, and specifically of this mild neurocognitive disorder, is crucial for a window of intervention prior to dementia. The investigators propose to evaluate a tablet version of a manual dexterity test that the investigators have already been able to test, in combination with assessments already established in the clinic and physiological data collected by a connected watch, to help diagnose neurocognitive disorders by confronting them with the clinical data that are the reference.

The investigators propose this multicenter observational study with a diagnostic aim. The study will involve 150 elderly people consulting one of the two participating memory centers. Three groups will be formed: 50 people with no cognitive dysfunction, 50 with a mild neurocognitive disorder, and 50 with a major neurocognitive disorder linked to Alzheimer's disease. These groups will be formed on the basis of the reference diagnosis established by the memory consultation teams, and the results of the patient's neuropsychological and medical assessments. The investigators will retrieve data from the medical record to classify cognitive status.

ELIGIBILITY:
Inclusion Criteria:

* elderly people consulting the memory center ;
* people with one of three documented cognitive diagnoses:
* major neurocognitive impairment due to Alzheimer's disease according to DSM-5 criteria,
* mild neurocognitive impairment
* no documented cognitive dysfunction after assessment at the memory center,
* willingness to participate in the study and sign the consent form.

Exclusion Criteria:

* persons with an illness affecting the hand (orthopedic, neurological, Parkinson's disease) that prevents them from using a touch-sensitive tablet;
* persons with other illnesses that may be responsible for loss of cognitive function (cerebrovascular disease, other neurological illnesses, psychiatric illnesses);
* persons benefiting from legal protection.

Ages: 60 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-04-17 (Estimated); Study Completion 2024-04-17 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, accuracy | through study completion, an average of 1 year
  Sensitivity, specificity, accuracy of the classification proposed by the algorithm in relation to the reference diagnosis.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Privé Gériatrique Les Magnolias, Ballainvilliers, Essonne
  - Hôpital Charles Foix, Ivry-sur-Seine, Val De Marne

IPD SHARING:
Plan to Share IPD: No
Personal data is password-protected and not shared; only investigators have access to this data. Study data that is shared is pseudonymized by a unique alphanumeric code generated by the application.